CLINICAL TRIAL: NCT03345927
Title: Investigation of Association Between Plasma S-adenosylhomocysteine Levels and Endothelial Dysfunction in Cardiovascular Disease Patients
Brief Title: Plasma S-adenosylhomocysteine Levels and Endothelial Dysfunction
Status: Completed | Type: Observational
Sponsor: Shenzhen Center for Disease Control and Prevention (Other Government)
Collaborators: Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Yunjun Xiao, Principal Investigator, Shenzhen Center for Disease Control and Prevention
Other Study IDs: ShenzhenCDC
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases
Keywords: S-adenosylhomocysteine; Endothelial function
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 10mL plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high cardiovascular risk group: no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To investigate the relationship betweeen plasma S-adenosylhomocysteine (SAH) levels and endothelial dysfunction, we plan to enroll approximately 150 patients with high risk of cardiovascualr disease,who will be measaured the flow-mediated dilation by B-ultrasound, and then measaured the plasma levels of methionine metabolites, such as SAH, SAM, and analyze the association.

DETAILED DESCRIPTION:
To investigate the relationship betweeen plasma S-adenosylhomocysteine (SAH) levels and endothelial dysfunction, we plan to enroll approximately 150 patients with high risk of cardiovascualr disease,who will be measaured the flow-mediated dilation by B-ultrasound, and then use HPLC-MS/MS to measaure the plasma levels of methionine metabolites, such as SAH, SAM, and use methylated specifical PCR to detect the promoter DNA methylation of p66shc, and use ELISA kits to measure the plasma ROS levels of CVD patients, such as MDA, 8-iso-prostaglandin F2a, and finally analyze the association between SAH, ROS levels, promoter DNA methylation of p66shc, and flow-mediated dilation.

ELIGIBILITY:
Inclusion Criteria:

* patients who have stable clinical conditions, except for acute coronary syndromes, and the availability of measurement of flow-mediated dilation, or have more than three cardiovascular traditional risk factors, such as smoking, alcohol use, obesity, hypertesion, diabetes, family history, and so on.

Exclusion Criteria:

* critical illness or hemodynamic instability other than acute coronary syndromes, surgery, or trauma within the previous month, known cancer, hepatic failure or hepatitis, or the use of drugs, such as anticancer agents, which would affect plasma tHcy concen-trations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with high cardiovascular risk, or diagnosed as coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Endothelial function | one month after enrollment
  measurement of flow-mediated dilation by B ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Yuebin Ke, Dr., Study Director — Shenzhen CDC
Locations (1):
- Chun Wang, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xiao Y, Xia J, Cheng J, Huang H, Zhou Y, Yang X, Su X, Ke Y, Ling W. Inhibition of S-Adenosylhomocysteine Hydrolase Induces Endothelial Dysfunction via Epigenetic Regulation of p66shc-Mediated Oxidative Stress Pathway. Circulation. 2019 May 7;139(19):2260-2277. doi: 10.1161/CIRCULATIONAHA.118.036336. PMID 30773021